CLINICAL TRIAL: NCT06105801
Title: A Multicenter Randomized Trial of EBUS-TBNA Versus Transbronchial Mediastinal Cryobiopsy for Adequacy of Next Generation Sequencing
Brief Title: EBUS-TBNA vs Transbronchial Mediastinal Cryobiopsy for Adequacy of Next Generation Sequencing
Acronym: FROSTBITE-3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Northwestern Medicine (Other); Johns Hopkins University (Other); Duke University (Other); Medical University of South Carolina (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Fabien Maldonado, Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: VICC-VDTHO23177; NCI-2023-08954 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBUS-TBNA Group (Active Comparator): The same needle gauge will be used for these participant to acquire the initial diagnosis on ROSE (either 21 or 22G). Using standard sampling techniques, the mass or LN will be penetrated with the needle as confirmed by ultrasound, and the needle will be passed back from the proximal to the distal ends of the node to obtain the samples for an adequate cell block.
  Interventions: Procedure: Endobronchial ultrasound with transbronchial needle aspiration; Procedure: Bronchoscopy
- Transbronchial Mediastinal Cryobiopsy Group (Experimental): The operator will switch to a flexible, single-use, 1.1 mm cryoprobe (Erbe 20402-401, Erbe, Tübingen, Germany) for these participants to obtain cryobiopsies. The operator will introduce the probe into the working channel of the EBUS bronchoscope. The cryoprobe will then be advanced toward the puncture site and inserted gently through the previous puncture site created by the initial EBUS-TBNA needle. The operator will confirm the placement of the probe via the EBUS image, and photo capture will be done. The cryo-probe will be activated and cooled for 3 seconds before retracting with the bronchoscope with the frozen biopsy tissue attached to the tip.
  Interventions: Procedure: Endobronchial ultrasound with transbronchial needle aspiration; Procedure: Bronchoscopy; Procedure: Cryobiopsy

INTERVENTIONS:
Procedure: Endobronchial ultrasound with transbronchial needle aspiration — Participants will undergo Endobronchial ultrasound with transbronchial needle aspiration
Procedure: Bronchoscopy — Participants will undergo Bronchoscopy
Procedure: Cryobiopsy — Participants will undergo Cryobiopsy
  Arms: Transbronchial Mediastinal Cryobiopsy Group

SUMMARY:
This is a multi-center clinical trial evaluating the effect of transbronchial mediastinal cryobiopsy for its ability to improve the likelihood of obtaining tissue sufficient for molecular analysis. Patients in outpatient clinics or pre-operative holding areas planning to undergo a bronchoscopic biopsy of a suspected malignant lesion (peripheral or mediastinal) for initial diagnosis, staging, or tissue acquisition for molecular analysis will be considered for enrollment and consented. Patients will only be enrolled if intraoperative ROSE suggests malignancy. Patients will be randomized to continue with the operator's initial EBUS-TBNA needle or switch to a cryoprobe to perform a sampling.

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate the utility of transbronchial mediastinal cryobiopsy on its ability to improve the likelihood of acquiring tissue sufficient for next-generation sequencing (NGS).

Safety Endpoints:

* Pneumothorax within 7 days of procedure
* Moderate bleeding defined as controlled with bronchoscope, saline, or epinephrine
* Serious bleeding is defined as uncontrolled, leading to respiratory failure, need for transfusion, or cardiovascular instability
* Respiratory failure is defined as a new oxygen requirement or escalation in oxygen delivery within 7 days of procedure
* Unplanned hospitalization related to the procedure within 7 days of procedure
* Death

Exploratory Endpoints:

* The proportion of samples adequate for NGS testing
* The proportion of samples with adequate PD-1 / PD-L1 immunohistochemical staining
* Proportion of samples that are adequate for complete NGS library sequencing
* Estimated total number of tumor cells per H&E-stained slide
* Histological disease subtyping

ELIGIBILITY:
Inclusion Criteria:

* Lesions on PET or CT concerning for primary or metastatic malignancy that are amenable to biopsy by linear EBUS
* Malignant cells present on rapid on-site cytological evaluation (ROSE)

Exclusion Criteria:

* Patient is known to be less than 18 years old
* Patient is known to be pregnant
* Patient is known to be a prisoner
* Operator deems lesion is not safe to biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of samples sufficient for next-generation sequencing testing | Up to 12 months
  Comparison of samples between arms that meet sufficiency criteria for NGS

SECONDARY OUTCOMES:
Proportion of samples with adequate PD-1 / PD-L1 immunohistochemical staining | Up to 12 months
  Comparison of samples between arms that meet PD-1/PD-L1 adequacy
Proportion of samples that are adequate for complete NGS library sequencing | Up to 12 months
  Comparison of samples between arms that meet sufficiency criteria and then are adequate for complete NGS library sequencing
Estimated total number of tumor cells per H&E-stained slide | Up to 12 Months
  Comparison of samples between arms of estimated tumor cells per H&E-stained field
Histological disease subtyping | Up to 12 Months
  Comparison of samples between arms for subtypes of lung malignancies (primary or metastatic)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Maldonado, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT06105801/ICF_000.pdf